CLINICAL TRIAL: NCT07103512
Title: Additional Effects of Scalene Hold Relax Technique With Conventional Physical Therapy On Pulmonary Function in Asthma Patient
Brief Title: Scalene Hold Relax Technique With Conventional Physical Therapy in Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/02186 Ayesha Sabir
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalene Hold Relax Technique (Experimental): Scalene Hold Relax Technique Scalene Hold for 10 Second 10 Repetition. Hold your arms behind your back to keep them from rising then slowly tilt your head trying to touch your ear to your shoulder. Bend your neck only as far as it is comfortable, and hold for 5 to 10 seconds. Relax your neck and repeat 2-3 times on each side. The treatment will be provided for 1-4 weeks as per need
  Interventions: Other: Scalene Hold Relax Technique
- Conventional physical Therapy (Active Comparator): Diaphragmatic Breathing Exercise Inhale through nose about 4 Seconds, hold Breath for 2 Seconds, repeat 5 times, exercise repeated for 2-3 days per week followed up to 4 weeks.
  + Buteyko Breathing Exercise Exhale slowly and then hold that breath. Use index figure and thumb to plug nose hold that breath until there is an urge to breathe and then inhale Breathe normally at least 10 second repeat several. Frequency 2-3 days per week with Moderate Intensity follow-up to 4weeks
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Scalene Hold Relax Technique — Scalene Hold Relax Technique Scalene Hold for 10 Second 10 Repetition. Hold your arms behind your back to keep them from rising then slowly tilt your head trying to touch your ear to your shoulder. Bend your neck only as far as it is comfortable, and hold for 5 to 10 seconds. Relax your neck and repeat 2-3 times on each side. The treatment will be provided for 1-4 weeks as per need
  Arms: Scalene Hold Relax Technique
Other: Conventional Physical Therapy — Diaphragmatic Breathing Exercise Inhale through nose about 4 Seconds, hold Breath for 2 Seconds, repeat 5 times, exercise repeated for 2-3 days per week followed up to 4 weeks.
  + Buteyko Breathing Exercise Exhale slowly and then hold that breath. Use index figure and thumb to plug nose hold that breath until there is an urge to breathe and then inhale Breathe normally at least 10 second repeat several. Frequency 2-3 days per week with Moderate Intensity follow-up to 4weeks
  Arms: Conventional physical Therapy

SUMMARY:
To determine the additional effects of scalene hold relax technique with conventional exercises on pulmonary function in asthma patients

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Allergic asthma
* Both male and female will be included
* Age between 20 to 44 years.

Exclusion Criteria:

* Patient who do not provide consent
* Patient with any comorbid condition such as cardiovascular disease diabetes or other chronic illness
* Patient with any psychological condition that may interfere with participation or adherence to the study protocol

Ages: 22 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | 4 week
  A simple questionnaire Objective to measure the adequacy of asthma control and change in asthma control which occur either spontaneously or as a result of treatment ACQ has multidimensional construct assessing symptoms (5 items -self-administering and rescue in bronchodilator use (1 item-self-administered and FEV1%(1 item completed by clinic staff Test Retest reproducibility Reported with high intraclass correlation coefficient =0.90 Internal Consistency yes 7 point scale (0=no impairment =6 maximum impairment for symptoms and rescue use and 7categories for FEV1%) Minimally imp difference Change in score 0.5 7 items (score Range 0 (Totally controlled and 6 Severely Uncontrolled)
Asthma Control Test | 4 week
  A patient self-administered tool for identifying those with poorly controlled asthma assess the frequency of shortness of breath and general asthma The Score Range from 5 (poor control of asthma) to 25 complete control of asthma) with higher scores reflecting greater asthma control. 5 items with 4-week recall on symptoms and daily functioning 5-point scale for symptom and activities 1=not controlled at all 5= completely controlled
Lara Asthma Symptoms Scale | 4 week
  The Lara Asthma Symptom Scale (LASS) is a validated tool designed to assess asthma symptoms in adults. It comprises eight questions that evaluate the frequency of various asthma-related symptoms over the past four weeks. Each question is scored on a 5-point Likert scale, where higher scores indicate more frequent symptoms. To interpret the LASS, sum the scores from all eight questions to obtain a total score ranging from 0 to 32. Higher total scores indicate more frequent and severe asthma symptoms, suggesting poorer asthma control.
FEV1 | 4 week
  Forced Expiratory Volume in 1 second, is a measurement of how much air a person can forcefully exhale from their lungs in one second.
FVC | 4 week
  Forced Vital Capacity, is a measurement of lung function assessed during spirometry. t represents the maximum amount of air that can be forcefully exhaled after a full inhalation.
PEF | 4 week
  Peak Expiratory Flow) spirometer, often a simple peak flow meter, is a device used to measure the speed of air exhaled from the lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Mānsehra, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No